CLINICAL TRIAL: NCT06735469
Title: Leveraging Discrete Choice Experiments to Increase Participant Diversity in Future Clinical Trials
Brief Title: Clinical Trial Preference Study
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Melissa M. Crane, PhD, Assistant Professor, Rush University Medical Center
Other Study IDs: ORA# 24021303; R03DK139135 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-12-16 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Clinical Trials

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Discrete choice experiment — Participants will state their preferences for 1) return of full versus limited results to participants (trust/personal benefit), 2) balancing a study's participant burden with the study's ability to address multiple research aims (burden/knowledge generation), 3) incentivizing clinical assessments vs. conducting home-based assessments (personal benefit/burden), and 4) results generalizable to specific social groups versus the broader population. Participants will evaluate these attributes within a hypothetical trial to prevent chronic diseases.

SUMMARY:
Population subgroups experiencing health disparities are often also underrepresented in clinical trials. These groups include individuals from minoritized racial and ethnic groups, people from lower socioeconomic backgrounds, and men or women, depending on the study area. Identifying approaches to reduce health disparities will remain stalled until clinical trials can recruit and retain diverse clinical trial participants. To improve recruitment across studies, there is a need to understand how diverse populations view specific clinical trial attributes that could be manipulated to increase interest in trials. To address this need, this project will use a discrete choice experiment to identify and prioritize specific trial attributes under investigators' control that could be leveraged to enhance clinical trial participation rates in underrepresented groups. This project will evaluate participants' preferences of 1) return of full versus limited results to participants, 2) balancing a study's participant burden with its ability to address multiple research aims, 3) incentivizing clinical assessments vs. conducting homebased assessments, and 4) results generalizable to specific social groups versus the broader population. This experiment will be conducted with a sample of potential clinical trial participants (N = 800) that is diverse in terms of self-reported gender, racial and ethnic identity, education, and chronic disease status. The results of this study will be used to design a randomized comparison of enhanced clinical trial attributes across multiple health conditions to evaluate whether using the enhanced trial features can more efficiently recruit underrepresented participants into clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Internet access with audio and visual capabilities
* Reside within the United States
* Read and speak English

Exclusion Criteria:

* Under 18 years of age
* No internet access
* Reside outside of the United States
* Do not read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: United States adults
Sampling Method: Non-Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Participant preference for clinical trial attributes | Baseline
  Utility values generated from multinomal logit estimates from a discrete choice experiment of 8 hypothetical choices (Trial A, B, or neither).

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available in the Open Science Framework. Data will be made available as soon as possible after the data collection period has ended and will occur after the study investigators have had reasonable time to prepare manuscripts.